CLINICAL TRIAL: NCT00591500
Title: A Model for Genetic Susceptibility: Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of New Mexico (Other); University of North Carolina (Other); University of Michigan (Other); University of California, Irvine (Other); New South Wales Cancer Control (Unknown); University of Tasmania (Other); Registro dei Tumori, Torino, Italy (Unknown); British Columbia Cancer Agency (Other); Cancer Care Ontario (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 99-087; CA83180
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Skin Cancer
Keywords: Melanoma; Skin cancer; Genetic Susceptibility; polymorphisms
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Genetic Predisposition to Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buccal swabs tissue

GROUPS / COHORTS (2):
- Control: The control group comprises patients with a first primary melanoma diagnosed in a twelve-month period.
  Interventions: Behavioral: Questionnaire
- Cases: Cases are patients diagnosed with a second or higher order primary in a six-year period.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Exposures of interest will be measured by a self-administered personal residence, occupation and vacation calendar, a telephone interview, and by testing DNA from buccal cells and blood, when available. Standardization of diagnosis will be undertaken by review of tissue slides. Questionnaire data will be completed by interviewers. DNA will be obtained from each individual in the form of 4-6 buccal swabs
  Groups: Control
Behavioral: Questionnaire — Exposures of interest will be measured by a self-administered personal residence, occupation and vacation calendar, a telephone interview, and by testing DNA from buccal cells and blood, when available. Standardization of diagnosis will be undertaken by review of tissue slides. Questionnaire data will be completed by interviewers. DNA will be obtained from each individual in the form of 4-6 buccal swabs.
  Groups: Cases

SUMMARY:
The goal of this study is to find out if some people are more likely to get melanoma, a form of skin cancer, than others are. To do this we will compare people who have had more than one melanoma to people who have had only one melanoma and to people who are similar but who have not developed melanoma.

People respond to the environment in different ways. Some may be born with genes that make them more likely to get this type of skin cancer. Each person has many ways to repair normal damage to their genes. Specific genes may affect the repair of sun damage. Other genes affect the way the skin itself reacts to the sun. We want to find out which genes have normal changes in them and lead to different responses to exposures, such as the sun. We also want to find out if sun habits are related to the way these genes work.

DETAILED DESCRIPTION:
The purpose of this study is to better understand genetic susceptibility to melanoma and the interactions of specific polymorphisms with each other and with environmental factors.

To accomplish this, buccal swabs or blood specimens from patients with melanoma (either single primary or multiple primary) have been collected. Specimens will be prepared in the Epidemiology Laboratory at MSKCC. They will be analyzed at MSKCC for INK4A (and functional assays for DNA repair capacity when blood is available) and the melanocortin gene (MC1R), at the University of North Carolina for polymorphisms in DNA repair genes and immune function genes, at the University of Pennsylvania for polymorphisms in the melanocortin receptor gene (MC1R) and immune function genes, and at the University of California (Irvine) for polymorphisms in metabolizing genes (P450's and GST's). Samples will be banked at MSKCC and the University of New Mexico. In order to perform this study, subjects from population-based registries in the United States (New Jersey, North Carolina, Michigan, San Diego/Imperial Counties), Canada (Cancer Care Ontario, British Columbia), Italy (Turin), Australia (New South Wales, Tasmania), were interviewed, asked to provide blood or buccal swab samples and asked to provide permission to obtain and review slides of their primary melanoma. This study is now closed to accrual.

ELIGIBILITY:
Inclusion Criteria:

- The subject must have a histologically confirmed invasive first primary melanoma newly diagnosed between January 1, 2000 and December 31, 2000.

OR the subject must have a histologically confirmed invasive or in situ second primary melanoma newly diagnosed between January 1, 1998 and December 31, 2003. One of the earlier primaries must be invasive melanoma OR the subject must be a randomly ascertained control from the general.

- The patient must be a resident of a one of the specific geographic areas participating in this study.

Exclusion Criteria:

* Subjects who do not speak English or Italian
* Subject is unable to sign informed consent
* Subject is unable to participate in telephone interview

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population-based registries in the United States
Sampling Method: Non-Probability Sample
Enrollment: 4082 (Actual)
Dates: Start 1999-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of INK4A and CDK4 mutation status and DNA repair gene, metabolizing gene, immune function gene, and melanocortin receptor gene polymorphism status; Interactions between polymorphisms and sun exposure history; Interactions among polymorphisms. | 2 years

SECONDARY OUTCOMES:
to examine psychosocial factors that predict skin cancer prevention behaviors including: participants' perceptions of future cancer risk, worry about cancer, self-efficacy, response-efficacy, and presence of family discussions about skin cancer risk. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Orlow, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering web site — http://www.mskcc.org